CLINICAL TRIAL: NCT02063464
Title: Collection of Blood From Patients With Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Blood Collection From People With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140056; 14-C-0056
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Cancer; Cancer of the Ovary; Ovarian Neoplasms
Keywords: Monocytes; Interferons Alpha and Gamma; tumoricidal; Natural History
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects w/ovarian, primary peritoneal or fallopian tube ca who are not currently on therapy and are screening for trials, being seen in consultation, or presenting for enrollment on a trial.

SUMMARY:
Background:

* Monocytes are a type of white blood cell found in human blood. They help the immune system. Researchers have found that monocytes taken from the blood of healthy people can kill tumor cells. Now they want to know if monocytes taken from the blood of people with ovarian cancer can kill tumor cells.
* In addition, native host anti-tumor cell mediated immune mechanisms may play a role in clinical outcome of epithelial ovarian cancer; data indicate that the presence of intra-tumoral CD3+ T-cells was shown to prognosticate improved outcome in advanced ovarian cancer. Furthermore, non-cellular components in the blood, such as exosomes, may influence outcome.

Objective:

- To see if monocytes taken from the blood of people with ovarian cancer can kill tumor cells.

Eligibility:

- Women 18 years and older with ovarian cancer.

Design:

* Participants will be screened with:
* Medical history and physical exam.
* Blood tests.
* CT scan of the chest, abdomen, and pelvis and/or an MRI. For these scans, they will lie in a machine that takes pictures of their body.
* A small amount of blood (two tubes) will be collected by needle during one visit.

DETAILED DESCRIPTION:
Background:

Using both in vitro and in vivo assays we have shown that human monocytes primed with Interferons alpha and gamma are tumoricidal and are capable of killing a number of tumor cell lines and human tumors implanted into immunocompromised mice. We have shown that monocytes isolated through elutriation at the NIH blood bank and monocytes isolated from anticoagulated peripheral blood from healthy women from the NIH blood bank are equally capable of killing tumor cells. No data have been collected as to whether monocytes from patients with Ovarian, Primary Peritoneal, or Fallopian Tube Cancer have tumoricidal properties. In addition, native host anti-tumor cell mediated immune mechanisms may play a role in clinical outcome of epithelial ovarian cancer; data indicate that the presence of intra-tumoral CD3+ T-cells was shown to prognosticate improved outcome in advanced ovarian cancer. Furthermore, noncellular components in the blood, such as exosomes, may influence outcome.

Objectives:

To obtain blood samples from patients with ovarian, primary peritoneal or fallopian tube cancer.

Eligibility:

Females greater than or equal to 18 years of age with a prior diagnosis of ovarian, primary peritoneal or fallopian tube cancer seen in the Women s Cancer Clinic of the NCI. Patients must be able and willing to provide informed consent.

Design:

We will collect approximately 20 ml of peripheral blood at a single time point from patients with ovarian, primary peritoneal or fallopian tube cancer who are not currently on therapy and are screening for trials, being seen in consultation, or presenting for enrollment on a clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA
* Females greater than or equal to 18 years of age with histologically proven ovarian, primary peritoneal or fallopian tube cancer.
* Currently not on therapy. Must be at least 2 weeks from prior therapy.
* Ability and willingness to provide informed consent to participation.

EXCLUSION CRITERIA

- Children are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants w/ovarian, primary peritoneal or fallopian tube cancer who are screening for trials, being seen in consultation, or presenting for enrollment on a clinical trial at the NIH Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
To obtain blood samples from patients with ovarian, primary peritoneal or fallopian tube cancer | Single blood collection upon enrollment
  A collection of blood samples from patients with ovarian, primary peritoneal or fallopian tube cancer

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Annunziata, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0056.html